CLINICAL TRIAL: NCT05164159
Title: The Comparison of Hemodynamic Effects Between Remimazolam-remifentanil and Propofol-remifentanil in Patients Undergoing Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2021-1440
Record Dates: First submitted 2021-12-15; First posted 2021-12-20 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Acute Cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol group (Active Comparator): During induction, the propofol group starts the effect site concentration at 4.0 ng/ml with TCI and adjusts it to around 3.0 ~ 4.0 ng/ml after intubation to maintain an appropriate EEG-based depth of anesthesia.
  Interventions: Drug: propofol group
- remimazolam group (Experimental): Arm Description: In the remimazolam group, start remimazolam at 6 mg/kg/hr and adjust it to 1 mg/kg/hr after loss of consciousness to maintain an appropriate EEG-based depth of anesthesia.
  Interventions: Drug: remimazolam group

INTERVENTIONS:
Drug: propofol group — During induction, the propofol group starts the effect site concentration at 4.0 ng/ml with TCI and adjusts it to around 3.0 ~ 4.0 ng/ml after intubation to maintain an appropriate EEG-based depth of anesthesia.
  Arms: propofol group
Drug: remimazolam group — In the remimazolam group, start remimazolam at 6 mg/kg/hr and adjust it to 1 mg/kg/hr after loss of consciousness to maintain an appropriate EEG-based depth of anesthesia.
  Arms: remimazolam group

SUMMARY:
This study is conducted to determine whether the occurrence of hypotension is reduced by the combined use of remimazolam and remifentanil compared to the conventional combination use of propofol and remifentanil. Patients enrolled in the study are infused continuously with either propofol or remimazolam from the start of anesthesia to the end of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. patients 19 years of age or older
2. the American Society of Anesthesiologists classification 1-3
3. patients undergoing laparoscopic cholecystectomy at Severance Hospital

Exclusion Criteria:

1. Emergency surgery,
2. patients with heart disease or arrhythmias,
3. patients undergoing concurrent surgery other than laparoscopic cholecystectomy,
4. obesity (BMI>30),
5. patients who were admitted on the surgery day,
6. foreigners,
7. illiteracy

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Percent of patients with hypotension event | from start of drugs to end of anesthesia on the surgery 1 day

SECONDARY OUTCOMES:
time-weighted average of hypotension | from start of drugs to end of anesthesia on the surgery 1 day
  time-weighted average of hypotension is calculated as the depth of hypotension below a MAP of 65 mm Hg (in millimeters of mercury) × time spent below a MAP of 65 mm Hg (in minutes) divided by total duration of operation (in minutes).
dose of Norepinephrine or nicardipine | from start of drugs to end of anesthesia on the surgery 1 day
difference of QOR-40 score | Baseline (preoperative period) and Postoperative day 1
  QoR-40 was developed by Myles et al and is a questionnaire that can examine the quality of recovery and health status of patients in the early postoperative period. Patients will also fill out a questionnaire before surgery for comparison with postoperative scores.
Heart rate variability | from start of drugs to end of anesthesia on the surgery 1 day
  Heart rate variability is a relatively easy and non-invasive measurement method that reflects the level of balance between the sympathetic and parasympathetic nerves at every moment using EKG records.
Sedline(Psi) | from start of drugs to end of anesthesia on the surgery 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Nyeo Koo, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No